CLINICAL TRIAL: NCT05239871
Title: Indirect Ultrasonographic Findings Predicting Parametrial Involvement in Severe Deep Endometriosis
Brief Title: Indirect Ultrasonographic Findings for Parametrial Involvement in Deep Endometriosis
Status: Completed | Type: Observational
Sponsor: Simone Ferrero (Other)
Responsible Party: Sponsor-Investigator, Simone Ferrero, Principal Investigator, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Organization: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Other Study IDs: ULTRA-PARAMETRENDO I
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Endometriosis; Deep Endometriosis
Keywords: Parametrial endometriosis; Deep endometriosis; Transvaginal Ultrasound
MeSH Terms: conditions — Endometriosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with surgical diagnosis of parametrial endometriosis: This cohort will include patients with surgical diagnosis of parametrial endometriosis
  Interventions: Diagnostic Test: Ultrasound
- Women without surgical diagnosis of parametrial endometriosis: This cohort will include patients without surgical diagnosis of parametrial endometriosis
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Preoperative transvaginal/transabdominal ultrasonography done according to IDEA criteria.

SUMMARY:
This study evaluated the use of ultrasonographic findings as a first-line imaging tool to raise indirect suspicion of parametrial involvement in women suspected of having severe endometriosis (DE).

DETAILED DESCRIPTION:
Ultrasonographic findings will be conventionally divided in:

* concomitant DE nodules
* indirect DE signs

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected deep endometriosis undergoing surgical approach

Exclusion Criteria:

* patients with a previous surgical diagnosis of endometriosis
* pazients with radiological evidence of parametrial endometriosis
* patients who could not undergo transvaginal and/or transabdominal ultrasound for any technical reason

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with suspected deep endometriosis undergoing surgical approach in a third-level referral center for endometriosis between January 2021 and December 2021
Sampling Method: Non-Probability Sample
Enrollment: 1078 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with a surgical diagnosis of parametrial endometriosis | At surgery
Number of significant ultrasonographic concomitant DE nodules predicting surgical involvement | 1 week before surgical approach
Number of significant ultrasonographic indirect DE signs predicting surgical involvement | 1 week before surgical approach

CONTACTS AND LOCATIONS:
Locations (1):
- Ginecologia - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guerriero S, Martinez L, Gomez I, Pascual MA, Ajossa S, Pagliuca M, Alcazar JL. Diagnostic accuracy of transvaginal sonography for detecting parametrial involvement in women with deep endometriosis: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2021 Nov;58(5):669-676. doi: 10.1002/uog.23754. PMID 34358386
- [Result] Mabrouk M, Raimondo D, Arena A, Iodice R, Altieri M, Sutherland N, Salucci P, Moro E, Seracchioli R. Parametrial Endometriosis: The Occult Condition that Makes the Hard Harder. J Minim Invasive Gynecol. 2019 Jul-Aug;26(5):871-876. doi: 10.1016/j.jmig.2018.08.022. Epub 2018 Aug 31. PMID 30176361
- [Result] Ceccaroni M, Clarizia R, Roviglione G. Nerve-sparing Surgery for Deep Infiltrating Endometriosis: Laparoscopic Eradication of Deep Infiltrating Endometriosis with Rectal and Parametrial Resection According to the Negrar Method. J Minim Invasive Gynecol. 2020 Feb;27(2):263-264. doi: 10.1016/j.jmig.2019.09.002. Epub 2019 Sep 10. PMID 31518711
- [Result] Guerriero S, Condous G, van den Bosch T, Valentin L, Leone FP, Van Schoubroeck D, Exacoustos C, Installe AJ, Martins WP, Abrao MS, Hudelist G, Bazot M, Alcazar JL, Goncalves MO, Pascual MA, Ajossa S, Savelli L, Dunham R, Reid S, Menakaya U, Bourne T, Ferrero S, Leon M, Bignardi T, Holland T, Jurkovic D, Benacerraf B, Osuga Y, Somigliana E, Timmerman D. Systematic approach to sonographic evaluation of the pelvis in women with suspected endometriosis, including terms, definitions and measurements: a consensus opinion from the International Deep Endometriosis Analysis (IDEA) group. Ultrasound Obstet Gynecol. 2016 Sep;48(3):318-32. doi: 10.1002/uog.15955. Epub 2016 Jun 28. PMID 27349699
- [Derived] Barra F, Zorzi C, Albanese M, Stepniewska A, Deromemaj X, De Mitri P, Roviglione G, Clarizia R, Gustavino C, Ferrero S, Ceccaroni M. Ultrasonographic Findings Indirectly Predicting Parametrial Involvement in Patients with Deep Endometriosis: The ULTRA-PARAMETRENDO I Study. J Minim Invasive Gynecol. 2023 Jan;30(1):61-72. doi: 10.1016/j.jmig.2022.10.008. Epub 2022 Oct 29. PMID 36591808